CLINICAL TRIAL: NCT00938704
Title: Study to Compare the Efficacy and Safety of Two Non-Preserved Artificial Tears for the Treatment of Dry Eye Signs and Symptoms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MA-OPT-09-002
Record Dates: First submitted 2009-07-10; First posted 2009-07-14 (Estimated); Results first posted 2011-10-31 (Estimated); Last update posted 2011-10-31 (Estimated); Status verified 2011-09

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Carboxymethylcellulose Sodium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): carboxymethylcellulose 0.5%, glycerin 0.9%
  Interventions: Drug: carboxymethylcellulose 0.5% +glycerin 0.9%
- 2 (Active Comparator): sodium hyaluronate 0.18%
  Interventions: Drug: sodium hyaluronate 0.18%

INTERVENTIONS:
Drug: carboxymethylcellulose 0.5% +glycerin 0.9% — To open, twist and pull tab to remove. Instill study medication as needed, but at least one drop 3 times a day as instructed in the protocol and then discard the container.
  Other Names: Optive™ Sensitive
  Arms: 1
Drug: sodium hyaluronate 0.18% — To open, twist and pull tab to remove. Instill study medication as needed, but at least one drop 3 times a day as instructed in the protocol and then discard the container.
  Other Names: Vismed®
  Arms: 2

SUMMARY:
To compare the efficacy and safety of two non-preserved artificial tears, (carboxymethylcellulose 0.5%, + glycerin 0.9% vs. sodium hyaluronate 0.18%) eye drops for the treatment of the signs and symptoms of dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Current use of an artificial tear product at least 2 times per day (e.g. for relief of dry eye symptoms of dryness).
* Be likely to complete the entire course of study and to comply with appropriate instructions

Exclusion Criteria:

* Have undergone refractive surgery (e.g., cataract surgery, PRK, LASIK, or any surgery involving a limbal or corneal incision) within the last 12 months.
* Have uncontrolled systemic disease
* Are currently using, or have used within 14 days of study enrollment, any ocular medications other than artificial tears
* Have anticipated contact lens wear during the study
* Have an active ocular infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2009-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Ulm, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Carboxymethylcellulose 0.5%, Glycerin 0.9%: carboxymethylcellulose 0.5%, glycerin 0.9%
- Sodium Hyaluronate 0.18%: sodium hyaluronate 0.18%
Period: Overall Study
Arm/Group | Carboxymethylcellulose 0.5%, Glycerin 0.9% | Sodium Hyaluronate 0.18%
Started | 33 | 37
Completed | 33 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carboxymethylcellulose 0.5%, Glycerin 0.9% | Sodium Hyaluronate 0.18% | Total
Number analyzed (Participants) | 33 | 37 | 70
Age Continuous [Mean (Full Range); unit: years] | 54.386 [20.277 to 87.485] | 48.787 [18.942 to 84.482] | 51.5865 [18.942 to 87.485]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 28 | 51
  Male | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Ocular Surface Disease Index (OSDI) at Week 2
Description: Change from baseline in OSDI at Week 2. The OSDI consists of 12 questions measuring the presence of ocular symptoms. Each of the 12 questions is assessed using a 5-point scale (0=none of the time; 4=all of the time). The score is converted to a 0-100 score where 0 is best and 100 is worst. Higher OSDI scores are associated with greater severity. A negative number change from baseline indicates improvement.
Time Frame: Baseline, Week 2
Population: Intent-to-Treat (ITT). The ITT population consisted of all patients who started the study (randomized).
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Carboxymethylcellulose 0.5%, Glycerin 0.9% | Sodium Hyaluronate 0.18%
Number analyzed (Participants) | 33 | 37
Scores on a Scale
  Baseline | 56.06 (13.43) | 54.292 (13.100)
  Week 2 | -27.048 (17.87) | -28.303 (21.821)

2. Secondary Outcome: Change From Baseline in Tear Breakup Time (TBUT) at Week 2
Description: Change from baseline in TBUT at Week 2. TBUT is defined as the time required for dry spots to appear on the surface of the eye after blinking. The longer it takes, the more stable the tear film. A positive number change from baseline indicates improvement.
Time Frame: Baseline, Week 2
Population: Intent-to-Treat (ITT). The ITT population consisted of all patients who started the study (randomized).
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Carboxymethylcellulose 0.5%, Glycerin 0.9% | Sodium Hyaluronate 0.18%
Number analyzed (Participants) | 33 | 37
Seconds
  Baseline | 6.501 (1.73) | 5.914 (1.646)
  Week 2 | 2.919 (2.388) | 2.538 (2.923)

3. Secondary Outcome: Change From Baseline in Corneal Staining at Week 2
Description: Change from baseline in corneal staining at Week 2. Staining of the cornea following ocular administration of fluorescein dye was graded using a 6-point scale (0=no staining, 5=diffuse staining). The higher the grade score, the worse the dry eye severity. A negative number change from baseline indicates improvement.
Time Frame: Baseline, Week 2
Population: Intent-to-Treat (ITT). The ITT population consisted of all patients who started the study (randomized).
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Carboxymethylcellulose 0.5%, Glycerin 0.9% | Sodium Hyaluronate 0.18%
Number analyzed (Participants) | 33 | 37
Scores on a Scale
  Baseline | 1.818 (0.779) | 1.608 (0.936)
  Week 2 | -1.288 (0.718) | -1.23 (1.090)

4. Secondary Outcome: Change From Baseline in Conjunctival Staining (Temporal) at Week 2
Description: Change from baseline in conjunctival (temporal) staining at Week 2. Staining of the conjunctiva following ocular administration of lissamine green dye was graded using a 6-point scale (0=no staining, 5=diffuse staining). The higher the grade score, the worse the dry eye severity. A negative number change from baseline indicates improvement.
Time Frame: Baseline, Week 2
Population: Intent-to-Treat (ITT). The ITT population consisted of all patients who started the study (randomized).
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Carboxymethylcellulose 0.5%, Glycerin 0.9% | Sodium Hyaluronate 0.18%
Number analyzed (Participants) | 33 | 37
Scores on a Scale
  Baseline | 1.818 (0.950) | 1.919 (1.010)
  Week 2 | -1.152 (0.972) | -1.216 (1.084)

5. Secondary Outcome: Change From Baseline in Conjunctival Staining (Nasal) at Week 2
Description: Change from baseline in conjunctival staining (nasal) at Week 2. Staining of the conjunctiva following ocular administration of lissamine green dye was graded using a 6-point scale (0=no staining, 5=diffuse staining). The higher the grade score, the worse the dry eye severity. A negative number change from baseline indicates improvement.
Time Frame: Baseline, Week 2
Population: Intent-to-Treat (ITT). The ITT population consisted of all patients who started the study (randomized).
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Carboxymethylcellulose 0.5%, Glycerin 0.9% | Sodium Hyaluronate 0.18%
Number analyzed (Participants) | 33 | 37
Scores on a Scale
  Baseline | 1.758 (0.902) | 2.000 (0.913)
  Week 2 | -1.061 (0.899) | -1.459 (1.043)

ADVERSE EVENTS:
Arm/Group | Carboxymethylcellulose 0.5%, Glycerin 0.9% | Sodium Hyaluronate 0.18%
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/37
Other Adverse Events (participants affected / at risk) | 0/33 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.